CLINICAL TRIAL: NCT03379311
Title: A Phase 1b, Open-Label, Multiple Dose, Proof-of-Concept Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AK002 in Patients With Atopic Keratoconjunctivitis, Vernal Keratoconjunctivitis, and Perennial Allergic Conjunctivitis
Brief Title: A Study of AK002 in Patients With Atopic Keratoconjunctivitis, Vernal Keratoconjunctivitis, and Perennial Allergic Conjunctivitis
Acronym: KRONOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AK002-005
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Atopic Keratoconjunctivitis; Vernal Keratoconjunctivitis; Perennial Allergic Conjunctivitis
Keywords: AKC; PAC; VKC
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — AK002

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: AK002 — AK002 is a humanized non-fucosylated immunoglobulin G1 (IgG1) monoclonal antibody directed against Siglec-8, a member of the CD33-related family of sialic acid-binding, immunoglobulin-like lectins (Siglecs).

SUMMARY:
This is a Phase 1b, open-label, study to assess the effects of AK002, given as monthly intravenous infusion for 6 doses at up to 3 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Male or female aged ≥18 and ≤80 years at the time of signing the informed consent form
3. Confirmed diagnosis of AKC, VKC, or PAC and an average total ACS score of ≥15 calculated from all daily ACS questionnaires completed during the screening period (minimum of 14 daily ACS questionnaires must be completed). Total ACS score is the sum of itching, light sensitivity, eye pain, foreign body sensation, and watering symptom scores (and excludes atopic dermatitis, allergic asthma, and allergic rhinitis scores).
4. History of topical corticosteroid and/or systemic corticosteroid use for the treatment of allergic conjunctivitis (AKC, VKC, or PAC)
5. Stable dose(s) of allowed AKC, VKC, or PAC medication(s) during the 14 days prior to Day 1; and commitment to remaining on the same dose(s) of AKC, VKC, or PAC medication(s) for the entire duration of study participation (unless dose modification is due to unforeseen medical necessity) per Section 8.1 and Section 8.2.
6. Willing and able to comply with the study procedures and visit schedule, including follow-up visits
7. Negative Screening ova and parasite test
8. Female patients must be either post-menopausal for at least 1 year with FSH level >40 mIU/mL at Screening or surgically sterile (tubal ligation, hysterectomy or bilateral oophorectomy) for at least 3 months, or if of child-bearing potential, have a negative pregnancy test and agree to use dual methods of contraception, or abstain from sexual activity from Screening until the end of the study, or for 120 days following the last dose of study drug, whichever is longer.

Male patients with female partners of childbearing potential must agree to use a highly effective method of contraception from Screening until the end of the study or for 120 days following the last dose of study drug, whichever is longer. All fertile men with female partners of childbearing potential should be instructed to contact the Investigator immediately if they suspect their partner might be pregnant (e.g., missed or late menstrual period) at any time during study participation.

Exclusion Criteria:

1. Known hypersensitivity to any constituent of the study drug
2. Women who are pregnant, breastfeeding, or planning to become pregnant while participating in the study
3. Presence of abnormal laboratory values considered to be clinically significant by the Investigator
4. Any disease or condition (medical or surgical) which, in the opinion of the Investigator, would place the patient at increased risk
5. History of malignancy, exempting: carcinoma in situ in the cervix, early stage prostate cancer, non-melanoma skin cancers, or cancers that have been in remission for more than 5 years and are considered cured (except for breast cancer). All history of malignancy (including diagnosis, dates, and compliance with cancer screening recommendations) must be documented and certified by the Investigator.
6. Contact lens use within 48 hours prior to first AK002 dose
7. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to administration of study drug (or 90 days or 5 half-lives, whichever is longer, for biologic products)
8. Treatment with chemotherapy or radiotherapy in the preceding 6 months
9. Treatment for a clinically significant helminthic parasitic infection within 6 months of screening
10. Use during the 30 days before Screening (or 5 half-lives, whichever is longer) or use during the Screening period of topical decongestants, topical vasoconstrictors, topical calcineurin inhibitors, topical corticosteroids*, omalizumab, dupilumab, systemic immunosuppressive drugs, or systemic corticosteroids with a daily dose >10 mg prednisone or equivalent per Section 8.1 and Section 8.2

    *Topical corticosteroids for atopic dermatitis, corticosteroid nasal sprays for rhinitis, and inhaled corticosteroids for allergic asthma are allowed.
11. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of the study drug administration
12. Positive hepatitis serology results, except for vaccinated patients or patients with past but resolved hepatitis, at Screening
13. Positive HIV serology results at Screening
14. Known history of alcohol, drug, or other substance abuse or dependence
15. Any other reason that (in the opinion of the Investigator or Medical Monitor) makes the patient unsuitable for enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability by evaluating Clinical laboratory parameters and adverse events assessed using the CTCAE version 4.03 | Adverse events will be collected starting from the time of first study drug infusion and ending at Day 309 (±7 Days) or the ET Visit unless directed otherwise by Allakos

SECONDARY OUTCOMES:
To evaluate the pharmacodynamics of AK002 in patients with AKC, VKC, or PAC as measured by changes from baseline in absolute peripheral blood counts of eosinophils and basophils | Starting pre-dose on day -1 to day 309 or early term visit
To evaluate the pharmacodynamics of AK002 using the Allergic Conjunctivitis Symptom Questionnaire (ACS) | Throughout the study from screening to day 309 or early term visit
  To evaluate the pharmacodynamics of AK002 in patients with AKC, VKC, or PAC as measured by changes from baseline symptoms associated with AKC, VKC, or PAC as measured daily by a disease-specific patient questionnaire, the Allergic Conjunctivitis Symptom Questionnaire (ACS)

CONTACTS AND LOCATIONS:
Overall Officials: Quan D Nguyen, MD, MSc, Principal Investigator — Stanford University
Locations (8):
- United States (8):
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Riverside Clinical Research, Edgewater, Florida
  - University of Maryland, Department of Ophthalmology and Visual Sciences, Baltimore, Maryland
  - Ocular Immunology and Uveitis Foundation, Waltham, Massachusetts
  - Tauber Eye Center, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Metropolitan Eye Research and Surgery Institute, Palisades Park, New Jersey
  - UPMC Eye Center, Pittsburgh, Pennsylvania